CLINICAL TRIAL: NCT06364215
Title: Posterior Wall Substrate Modification Using Irreversible Electroporation for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Posterior Wall Substrate Modification Using Irreversible Electroporation for Paroxysmal Atrial Fibrillation
Acronym: (SMILE-AF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment related to ILR coverage barriers and the resulting inability to meet timelines with the available funding.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry); Databean (Industry)
Responsible Party: Principal Investigator, Jorge E. Romero, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P000883
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: pulsed field ablation; paroxysmal atrial fibrillation; left atrium posterior wall isolation; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pulmonary Vein Isolation (PVI) only (Active Comparator): Pulsed field ablation of the pulmonary veins only.
  Interventions: Device: Farapulse PFA, Pulmonary Vein Isolation alone
- Pulmonary Vein Isolation and Posterior Wall Isolation ( PVI+PWI) (Active Comparator): Pulsed field ablation of the pulmonary veins and the posterior wall of the left atrium.
  Interventions: Device: Farapulse PFA, Pulmonary Vein Isolation and Left atrial Posterior Wall Isolation

INTERVENTIONS:
Device: Farapulse PFA, Pulmonary Vein Isolation alone — Ablation of the pulmonary veins for the treatment of Paroxysmal Atrial Fibrillation using pulsed field ablation.
  Arms: Pulmonary Vein Isolation (PVI) only
Device: Farapulse PFA, Pulmonary Vein Isolation and Left atrial Posterior Wall Isolation — Ablation of the pulmonary veins and the left atrium posterior wall for the treatment of Paroxysmal Atrial Fibrillation using pulsed field ablation.
  Arms: Pulmonary Vein Isolation and Posterior Wall Isolation ( PVI+PWI)

SUMMARY:
The purpose of this study is to compare the efficacy and safety between pulmonary vein isolation (PVI) alone versus PVI with left atrial (LA) posterior wall isolation (PWI) using pulsed-field ablation (PFA) in the treatment of patients with paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, randomized, multi-center, Investigational Device Exemption (IDE) study. Subjects undergoing first-time ablation for paroxysmal atrial fibrillation will be randomized to receive either pulmonary vein isolation (PVI) alone or PVI combined with posterior wall isolation (PWI) using pulsed field ablation (PFA) with the FARAWAVE PFA catheter.

Following the index procedure, all participants will enter a 3-month blanking period, during which they will be closely monitored. After this period, anti-arrhythmic drug (AAD) therapy will be discontinued for all patients. Throughout the entire study, patients will be monitored using an implantable loop recorder (ILR) to assess the primary outcome of efficacy.

The study includes a 12-month follow-up period, and the primary objective is to assess and compare the efficacy, defined as an improvement in freedom from all-atrial arrhythmias, and safety, defined as the occurrence of all procedure-related complications.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age 21-90 years.
4. Symptomatic PAF whether failed AAD or not.
5. At least one symptomatic episode of PAF lasting <7 days, documented on electrocardiogram (ECG), Holter, ZioPatch, ILR, or smartwatch recording in the year prior to enrollment.
6. Patients undergoing first time ablation for AF.
7. Subject has any commercially available implantable loop recorder (ILR) or agrees to have one implanted prior or during the ablation procedure.

Exclusion Criteria:

1. Persistent atrial fibrillation (PeAF) (> 7 days in duration).
2. Atrial arrhythmias secondary to electrolyte imbalance, thyroid disease, or other reversible non-cardiac cause.
3. Previous surgical or catheter ablation of AF.
4. Previous valve surgery, ventriculotomy, atriotomy, or presence of a mitral mechanical prosthetic or bioprosthetic valve.
5. Left atrium anteroposterior (LA AP) diameter >55 mm or indexed left atrium (LA) volume >48 ml/m2.
6. Contraindications to oral or systemic anticoagulation.
7. Previous thromboembolic event (including ischemic strokes and TIA) within the last 3 months.
8. Previous myocardial infarction or percutaneous coronary intervention within the past 2 months.
9. Coronary Artery Bypass Grafting (CABG) surgery within the past 6 months (180 days).
10. Pregnancy.
11. History of PV stenosis.
12. History of severe pulmonary hypertension.
13. History of diaphragmatic paresis or hemi-paresis.
14. History of heart transplantation.
15. History of blood clotting or bleeding abnormalities.
16. Life expectancy of less than 12 months.
17. Presence of intracardiac thrombus.
18. Complex congenital heart disease, including tetralogy of Fallot, ventricular septal defects, Ebstein's anomaly, systemic right ventricle, and transposition of the great arteries.
19. Intracardiac or vascular abnormalities that preclude adequate catheter introduction or manipulation within the LA.
20. Pacing dependent patients.
21. Active malignancy or history of treated malignancy within 12 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma).
22. Active systemic infection.
23. Participation in any other AF-related randomized clinical trial.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Procedural success, defined as freedom from of all documented atrial arrhythmias episodes after the 3-month blanking period. | 12 months
  will be assessed by:
  * Occurrence of all atrial arrhythmias after the 3-month blanking period.
  * Any cardioversion for atrial fibrillation (AF), atrial flutter (AFL), or atrial tachycardia (AT) after the 3-month blanking period.
  * Use of any type I or type III antiarrhythmic medication for the treatment of AF, AFL, or AT after the 3-month blanking period, or the use of amiodarone at any time.
  * Re-ablation of AF, AFL, or AT.
The primary safety endpoint is a composite of acute procedure-related complications and any other major adverse events within the 12 months following the ablation procedure. | 12 Months
  All number of acute procedure-related complications will be reported and assessed including: atrio-esophageal fistula, cardiac perforation, pulmonary vein (PV) stenosis, acute kidney injury, phrenic nerve paralysis, thromboembolic events, stroke, or transient ischemic attacks (TIA), and other major adverse events within the 12 months following the ablation procedure: pericarditis cardiac tamponade pericardial effusion, coronary artery spasm, Vascular access complication/major bleeding, local hematoma, ecchymosis left atrium or vascular laceration

SECONDARY OUTCOMES:
Freedom from atrial arrhythmias medication | 12 Months
  Time and dose of anti arrhythmic medications use will be compared between the two groups.
Procedural time | 12 Months
  procedural time will be compared among groups.
Procedure-related Recurrencies | 12 Months
  Rate of PV and PW reconnection in patients undergoing repeat ablation procedures for recurrence of AF.
Atrial Fibrillation Effect on Quality-of-life Questionnaire (AFEQT). | 12 Months
  It reports scores from 0 to 100. A score of 0 corresponds to complete disability, while a score of 100 describes the highest level of QoL
Use of amiodarone | 12 months
  Number of patients using amiodarone, and duration of using it will be compared among groups.
Complications. | 12 Months.
  Incidence of acute procedure-related complications and long-term procedure-related complication.
fluoroscopy time. | during 1-2 hours procedure.
  fluoroscopy time will be asses between the two groups.
Pulsed field ablation (PFA) applications during procedure. | During 1-2 hours procedure.
  The PFA count will be compared by the two groups.
first-pass pulmonary vein isolation (PVI). | During 1-2 hours procedure.
  the rates of first pass PVI will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Romero, MD, Principal Investigator — Massachusetts General Hospital; William H Sauer, MD, Principal Investigator — Massachusetts General Hospital
Locations (18):
- United States (18):
  - Grandview Medical Center, Birmingham, Alabama
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Vincent's Health System, Inc. d/b/a Ascension St. Vincent's, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Corewell Health William Beaumont Hospital, Royal Oak, Michigan
  - The Valley Hospital, Paramus, New Jersey
  - North Shore University Hospital, Northwell Health, Manhasset, New York
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Orion Medical, Houston, Texas
  - Methodist Hospital-San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Rahman F, Kwan GF, Benjamin EJ. Global epidemiology of atrial fibrillation. Nat Rev Cardiol. 2016 Jul 14;13(8):501. doi: 10.1038/nrcardio.2016.114. No abstract available. PMID 27411521
- [Background] Wazni OM, Dandamudi G, Sood N, Hoyt R, Tyler J, Durrani S, Niebauer M, Makati K, Halperin B, Gauri A, Morales G, Shao M, Cerkvenik J, Kaplon RE, Nissen SE; STOP AF First Trial Investigators. Cryoballoon Ablation as Initial Therapy for Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):316-324. doi: 10.1056/NEJMoa2029554. Epub 2020 Nov 16. PMID 33197158
- [Background] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159
- [Background] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbuchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 1;383(14):1305-1316. doi: 10.1056/NEJMoa2019422. Epub 2020 Aug 29. PMID 32865375
- [Background] Chew DS, Jones KA, Loring Z, Black-Maier E, Noseworthy PA, Exner DV, Packer DL, Grant J, Mark DB, Piccini JP. Diagnosis-to-ablation time predicts recurrent atrial fibrillation and rehospitalization following catheter ablation. Heart Rhythm O2. 2021 Nov 19;3(1):23-31. doi: 10.1016/j.hroo.2021.11.012. eCollection 2022 Feb. PMID 35243432
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Romero J, Gabr M, Alviz I, Briceno D, Diaz JC, Rodriguez D, Patel K, Polanco D, Trivedi C, Mohanty S, Della Rocca D, Lakkireddy D, Natale A, Di Biase L. Focal impulse and rotor modulation guided ablation versus pulmonary vein isolation for atrial fibrillation: A meta-analysis of head-to-head comparative studies. J Cardiovasc Electrophysiol. 2021 Jul;32(7):1822-1832. doi: 10.1111/jce.15036. Epub 2021 May 27. PMID 33844385
- [Background] Atienza F, Almendral J, Jalife J, Zlochiver S, Ploutz-Snyder R, Torrecilla EG, Arenal A, Kalifa J, Fernandez-Aviles F, Berenfeld O. Real-time dominant frequency mapping and ablation of dominant frequency sites in atrial fibrillation with left-to-right frequency gradients predicts long-term maintenance of sinus rhythm. Heart Rhythm. 2009 Jan;6(1):33-40. doi: 10.1016/j.hrthm.2008.10.024. Epub 2008 Oct 22. PMID 19121797
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] Kistler PM, Chieng D, Sugumar H, Ling LH, Segan L, Azzopardi S, Al-Kaisey A, Parameswaran R, Anderson RD, Hawson J, Prabhu S, Voskoboinik A, Wong G, Morton JB, Pathik B, McLellan AJ, Lee G, Wong M, Finch S, Pathak RK, Raja DC, Sterns L, Ginks M, Reid CM, Sanders P, Kalman JM. Effect of Catheter Ablation Using Pulmonary Vein Isolation With vs Without Posterior Left Atrial Wall Isolation on Atrial Arrhythmia Recurrence in Patients With Persistent Atrial Fibrillation: The CAPLA Randomized Clinical Trial. JAMA. 2023 Jan 10;329(2):127-135. doi: 10.1001/jama.2022.23722. PMID 36625809
- [Background] Markman TM, Hyman MC, Kumareswaran R, Arkles JS, Santangeli P, Schaller RD, Supple GE, Frankel DS, Riley MP, Lin D, Garcia F, Dixit S, Callans DJ, Marchlinski FE, Nazarian S. Durability of posterior wall isolation after catheter ablation among patients with recurrent atrial fibrillation. Heart Rhythm. 2020 Oct;17(10):1740-1744. doi: 10.1016/j.hrthm.2020.05.005. Epub 2020 May 7. PMID 32389682
- [Background] Kumar P, Bamimore AM, Schwartz JD, Chung EH, Gehi AK, Kiser AC, Hummel JP, Mounsey JP. Challenges and Outcomes of Posterior Wall Isolation for Ablation of Atrial Fibrillation. J Am Heart Assoc. 2016 Sep 23;5(9):e003885. doi: 10.1161/JAHA.116.003885. PMID 27663412
- [Background] Aryana A, Thiemann AM, Pujara DK, Cossette LL, Allen SL, Bowers MR, Gandhavadi M, Heath R, Trivedi AD, O'Neill PG, Ellis ER, d'Avila A. Pulmonary Vein Isolation With and Without Posterior Wall Isolation in Paroxysmal Atrial Fibrillation: IMPPROVE-PAF Trial. JACC Clin Electrophysiol. 2023 May;9(5):628-637. doi: 10.1016/j.jacep.2023.01.014. Epub 2023 Mar 22. PMID 37225309
- [Background] Reddy VY, Anic A, Koruth J, Petru J, Funasako M, Minami K, Breskovic T, Sikiric I, Dukkipati SR, Kawamura I, Neuzil P. Pulsed Field Ablation in Patients With Persistent Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1068-1080. doi: 10.1016/j.jacc.2020.07.007. PMID 32854842
- [Background] Tovar O, Tung L. Electroporation of cardiac cell membranes with monophasic or biphasic rectangular pulses. Pacing Clin Electrophysiol. 1991 Nov;14(11 Pt 2):1887-92. doi: 10.1111/j.1540-8159.1991.tb02785.x. PMID 1721194
- [Background] Nikolski VP, Efimov IR. Electroporation of the heart. Europace. 2005 Sep;7 Suppl 2:146-54. doi: 10.1016/j.eupc.2005.04.011. PMID 16102512
- [Background] Fuller IA, Wood MA. Intramural coronary vasculature prevents transmural radiofrequency lesion formation: implications for linear ablation. Circulation. 2003 Apr 8;107(13):1797-803. doi: 10.1161/01.CIR.0000058705.97823.F4. Epub 2003 Mar 24. PMID 12665492
- [Background] Lavee J, Onik G, Mikus P, Rubinsky B. A novel nonthermal energy source for surgical epicardial atrial ablation: irreversible electroporation. Heart Surg Forum. 2007;10(2):E162-7. doi: 10.1532/HSF98.20061202. PMID 17597044
- [Background] Hong J, Stewart MT, Cheek DS, Francischelli DE, Kirchhof N. Cardiac ablation via electroporation. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:3381-4. doi: 10.1109/IEMBS.2009.5332816. PMID 19963798
- [Background] Wittkampf FH, van Driel VJ, van Wessel H, Vink A, Hof IE, Grundeman PF, Hauer RN, Loh P. Feasibility of electroporation for the creation of pulmonary vein ostial lesions. J Cardiovasc Electrophysiol. 2011 Mar;22(3):302-9. doi: 10.1111/j.1540-8167.2010.01863.x. PMID 20653809
- [Background] Wittkampf FH, van Driel VJ, van Wessel H, Neven KG, Grundeman PF, Vink A, Loh P, Doevendans PA. Myocardial lesion depth with circular electroporation ablation. Circ Arrhythm Electrophysiol. 2012 Jun 1;5(3):581-6. doi: 10.1161/CIRCEP.111.970079. Epub 2012 Apr 6. PMID 22492429
- [Background] Cochet H, Nakatani Y, Sridi-Cheniti S, Cheniti G, Ramirez FD, Nakashima T, Eggert C, Schneider C, Viswanathan R, Derval N, Duchateau J, Pambrun T, Chauvel R, Reddy VY, Montaudon M, Laurent F, Sacher F, Hocini M, Haissaguerre M, Jais P. Pulsed field ablation selectively spares the oesophagus during pulmonary vein isolation for atrial fibrillation. Europace. 2021 Sep 8;23(9):1391-1399. doi: 10.1093/europace/euab090. PMID 33961027
- [Background] Reddy VY, Koruth J, Jais P, Petru J, Timko F, Skalsky I, Hebeler R, Labrousse L, Barandon L, Kralovec S, Funosako M, Mannuva BB, Sediva L, Neuzil P. Ablation of Atrial Fibrillation With Pulsed Electric Fields: An Ultra-Rapid, Tissue-Selective Modality for Cardiac Ablation. JACC Clin Electrophysiol. 2018 Aug;4(8):987-995. doi: 10.1016/j.jacep.2018.04.005. Epub 2018 May 11. PMID 30139499
- [Background] Steiger NA, Romero JE. Pulsed-field ablation: What are the unknowns and when will they cease to concern us? J Cardiovasc Electrophysiol. 2022 Jul;33(7):1489-1493. doi: 10.1111/jce.15521. Epub 2022 May 25. No abstract available. PMID 35510406
- [Background] Stewart MT, Haines DE, Verma A, Kirchhof N, Barka N, Grassl E, Howard B. Intracardiac pulsed field ablation: Proof of feasibility in a chronic porcine model. Heart Rhythm. 2019 May;16(5):754-764. doi: 10.1016/j.hrthm.2018.10.030. Epub 2018 Oct 30. PMID 30385383
- [Background] Yavin H, Shapira-Daniels A, Barkagan M, Sroubek J, Shim D, Melidone R, Anter E. Pulsed Field Ablation Using a Lattice Electrode for Focal Energy Delivery: Biophysical Characterization, Lesion Durability, and Safety Evaluation. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e008580. doi: 10.1161/CIRCEP.120.008580. Epub 2020 May 6. PMID 32372696
- [Background] Koruth JS, Kuroki K, Kawamura I, Stoffregen WC, Dukkipati SR, Neuzil P, Reddy VY. Focal Pulsed Field Ablation for Pulmonary Vein Isolation and Linear Atrial Lesions: A Preclinical Assessment of Safety and Durability. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e008716. doi: 10.1161/CIRCEP.120.008716. Epub 2020 May 6. PMID 32370542
- [Background] Reddy VY, Anter E, Rackauskas G, Peichl P, Koruth JS, Petru J, Funasako M, Minami K, Natale A, Jais P, Nakagawa H, Marinskis G, Aidietis A, Kautzner J, Neuzil P. Lattice-Tip Focal Ablation Catheter That Toggles Between Radiofrequency and Pulsed Field Energy to Treat Atrial Fibrillation: A First-in-Human Trial. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e008718. doi: 10.1161/CIRCEP.120.008718. Epub 2020 May 8. PMID 32383391
- [Background] Loh P, van Es R, Groen MHA, Neven K, Kassenberg W, Wittkampf FHM, Doevendans PA. Pulmonary Vein Isolation With Single Pulse Irreversible Electroporation: A First in Human Study in 10 Patients With Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2020 Oct;13(10):e008192. doi: 10.1161/CIRCEP.119.008192. Epub 2020 Sep 8. PMID 32898450
- [Background] Tohoku S, Chun KRJ, Bordignon S, Chen S, Schaack D, Urbanek L, Ebrahimi R, Hirokami J, Bologna F, Schmidt B. Findings from repeat ablation using high-density mapping after pulmonary vein isolation with pulsed field ablation. Europace. 2023 Feb 16;25(2):433-440. doi: 10.1093/europace/euac211. PMID 36427201
- [Background] Kawamura I, Neuzil P, Shivamurthy P, Kuroki K, Lam J, Musikantow D, Chu E, Turagam MK, Minami K, Funasako M, Petru J, Choudry S, Miller MA, Langan MN, Whang W, Dukkipati SR, Koruth JS, Reddy VY. How does the level of pulmonary venous isolation compare between pulsed field ablation and thermal energy ablation (radiofrequency, cryo, or laser)? Europace. 2021 Nov 8;23(11):1757-1766. doi: 10.1093/europace/euab150. PMID 34151947
- [Background] Lee JM, Shim J, Park J, Yu HT, Kim TH, Park JK, Uhm JS, Kim JB, Joung B, Lee MH, Kim YH, Pak HN; POBI-AF Investigators. The Electrical Isolation of the Left Atrial Posterior Wall in Catheter Ablation of Persistent Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Nov;5(11):1253-1261. doi: 10.1016/j.jacep.2019.08.021. Epub 2019 Oct 30. PMID 31753429
- [Background] Aryana A, Allen SL, Pujara DK, Bowers MR, O'Neill PG, Yamauchi Y, Shigeta T, Vierra EC, Okishige K, Natale A. Concomitant Pulmonary Vein and Posterior Wall Isolation Using Cryoballoon With Adjunct Radiofrequency in Persistent Atrial Fibrillation. JACC Clin Electrophysiol. 2021 Feb;7(2):187-196. doi: 10.1016/j.jacep.2020.08.016. Epub 2020 Oct 28. PMID 33602399
- [Background] Ahn J, Shin DG, Han SJ, Lim HE. Does isolation of the left atrial posterior wall using cryoballoon ablation improve clinical outcomes in patients with persistent atrial fibrillation? A prospective randomized controlled trial. Europace. 2022 Jul 21;24(7):1093-1101. doi: 10.1093/europace/euac005. PMID 35138376
- [Background] Abhayaratna WP, Seward JB, Appleton CP, Douglas PS, Oh JK, Tajik AJ, Tsang TS. Left atrial size: physiologic determinants and clinical applications. J Am Coll Cardiol. 2006 Jun 20;47(12):2357-63. doi: 10.1016/j.jacc.2006.02.048. PMID 16781359
- [Background] Nattel S, Burstein B, Dobrev D. Atrial remodeling and atrial fibrillation: mechanisms and implications. Circ Arrhythm Electrophysiol. 2008 Apr;1(1):62-73. doi: 10.1161/CIRCEP.107.754564. No abstract available. PMID 19808395
- [Background] Lim HS, Hocini M, Dubois R, Denis A, Derval N, Zellerhoff S, Yamashita S, Berte B, Mahida S, Komatsu Y, Daly M, Jesel L, Pomier C, Meillet V, Amraoui S, Shah AJ, Cochet H, Sacher F, Jais P, Haissaguerre M. Complexity and Distribution of Drivers in Relation to Duration of Persistent Atrial Fibrillation. J Am Coll Cardiol. 2017 Mar 14;69(10):1257-1269. doi: 10.1016/j.jacc.2017.01.014. PMID 28279292
- [Background] Castiello T, Georgiopoulos G, Finocchiaro G, Claudia M, Gianatti A, Delialis D, Aimo A, Prasad S. COVID-19 and myocarditis: a systematic review and overview of current challenges. Heart Fail Rev. 2022 Jan;27(1):251-261. doi: 10.1007/s10741-021-10087-9. Epub 2021 Mar 24. PMID 33761041
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Huo Y, Gaspar T, Schonbauer R, Wojcik M, Fiedler L, Roithinger FX, Martinek M, Purerfellner H, Kirstein B, Richter U, Ulbrich S, Mayer J, Krahnefeld O, Agdirlioglu T, Zedda A, Piorkowski J, Piorkowski C. Low-Voltage Myocardium-Guided Ablation Trial of Persistent Atrial Fibrillation. NEJM Evid. 2022 Nov;1(11):EVIDoa2200141. doi: 10.1056/EVIDoa2200141. Epub 2022 Oct 19. PMID 38319851
- [Background] DeLurgio DB, Crossen KJ, Gill J, Blauth C, Oza SR, Magnano AR, Mostovych MA, Halkos ME, Tschopp DR, Kerendi F, Taigen TL, Shults CC, Shah MH, Rajendra AB, Osorio J, Silver JS, Hook BG, Gilligan DM, Calkins H. Hybrid Convergent Procedure for the Treatment of Persistent and Long-Standing Persistent Atrial Fibrillation: Results of CONVERGE Clinical Trial. Circ Arrhythm Electrophysiol. 2020 Dec;13(12):e009288. doi: 10.1161/CIRCEP.120.009288. Epub 2020 Nov 13. PMID 33185144
- [Background] Romero J, Polanco D, Gabr M, Alviz I, Diaz JC, Briceno D, Velasco A, Patel K, Natale A, Di Biase L. Posterior Wall Electrical Isolation in Patients Undergoing Catheter Ablation for Paroxysmal and Nonparoxysmal Atrial Fibrillation. JACC Clin Electrophysiol. 2023 Apr;9(4):583-585. doi: 10.1016/j.jacep.2022.11.007. Epub 2023 Jan 18. No abstract available. PMID 36752475
- [Background] Turagam MK, Neuzil P, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Lemoine MD, Ruwald M, Mulder BA, Rollin A, Lehrmann H, Fink T, Jurisic Z, Chaumont C, Adelino R, Nentwich K, Gunawardene M, Ouss A, Heeger CH, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Kueffer T, Rahe G, Reddy VY. Safety and Effectiveness of Pulsed Field Ablation to Treat Atrial Fibrillation: One-Year Outcomes From the MANIFEST-PF Registry. Circulation. 2023 Jul 4;148(1):35-46. doi: 10.1161/CIRCULATIONAHA.123.064959. Epub 2023 May 18. PMID 37199171
- [Background] Ekanem E, Reddy VY, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Rillig A, Mulder BA, Johannessen A, Rollin A, Lehrmann H, Sohns C, Jurisic Z, Savoure A, Combes S, Nentwich K, Gunawardene M, Ouss A, Kirstein B, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Turagam MK, Neuzil P; MANIFEST-PF Cooperative. Multi-national survey on the methods, efficacy, and safety on the post-approval clinical use of pulsed field ablation (MANIFEST-PF). Europace. 2022 Sep 1;24(8):1256-1266. doi: 10.1093/europace/euac050. PMID 35647644
- [Background] Mohanty S, Casella M, Compagnucci P, Torlapati PG, Della Rocca DG, La Fazia VM, Gianni C, Chierchia GB, MacDonald B, Mayedo A, Khan UN, Allison J, Bassiouny M, Gallinghouse GJ, Burkhardt JD, Horton R, Al-Ahmad A, Di Biase L, de Asmundis C, Russo AD, Natale A. Acute Kidney Injury Resulting From Hemoglobinuria After Pulsed-Field Ablation in Atrial Fibrillation: Is it Preventable? JACC Clin Electrophysiol. 2024 Apr;10(4):709-715. doi: 10.1016/j.jacep.2023.12.008. Epub 2024 Feb 1. PMID 38310489
- [Background] Venier S, Vaxelaire N, Jacon P, Carabelli A, Desbiolles A, Garban F, Defaye P. Severe acute kidney injury related to haemolysis after pulsed field ablation for atrial fibrillation. Europace. 2023 Dec 28;26(1):euad371. doi: 10.1093/europace/euad371. PMID 38175788